CLINICAL TRIAL: NCT00664170
Title: A Bioequivalence Study of Docetaxel for Injectable Emulsion (ANX-514) in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mast Therapeutics, Inc. (Industry)
Responsible Party: Michele Yelmene, Adventrx Pharmaceuticals, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ANX 514-01
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2009-05-28 (Estimated); Status verified 2009-05

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): ANX-514
  Interventions: Drug: ANX-514
- 2 (Active Comparator): Taxotere
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: ANX-514 — 75 mg/m^2
  Other Names: Docetaxel for Injectable Emulsion
  Arms: 1
Drug: docetaxel — 75 mg/m^2
  Other Names: Taxotere
  Arms: 2

SUMMARY:
The purpose of this study is to compare an injectable emulsion form of docetaxel to Taxotere in patients with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old.
* Advanced cancer potentially sensitive to single agent docetaxel; ie.. locally advanced or metastatic breast cancer, locally advanced non-small cell lung cancer, hormone refractory metastatic prostate cancer, other tumor type with no standard treatment.
* ECOG performance status of 0-2 and Karnofsky Score of 100-70.

Exclusion Criteria:

* Patients who have more effective therapy available than single agent docetaxel for the malignancy.
* Pregnancy or lactation.
* Intolerance to any antineoplastic agents belonging to the taxoid family.
* Hypersensitivity to drugs formulated with polysorbate 80.
* Active infection.
* Prior anticancer therapy within 30 days prior to the first day of study treatment.
* Participation in another experimental drug study within 30 days prior to the first day of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic equivalence of ANX-514 and Taxotere

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Stewart, MBA, Study Director — Mast Therapeutics, Inc.
Locations (13):
- United States (3):
  - Northwest Alabama Cancer Center, Muscle Shoals, Alabama
  - UCSD Moores Cancer Center, La Jolla, California
  - Signal Point Hematology/Oncology Inc., Middletown, Ohio
- Argentina (8):
  - Hospital Universitario Austral, Buenos Aires, Buenos Aires
  - Centro Oncologico de Rosario, Rosario, Santa Fe Province
  - Hospital Regional de Concepcion, Concepción, Tucumán Province
  - Marcelo T de Alvear, Buenos Aires
  - Centro Oncologico de Integracion Regional, Mendoza
  - Hospital Privado Santa Clara de Asis, Salta
  - Centro Medico San Roque, San Miguel de Tucumán
  - Isis Centro Especializado, Santa Fe
- Estonia (2):
  - Tallinn Cancer Clinic, Tallinn
  - Tartu University Hospital, Clinic of Hematology and Oncology, Tartu